CLINICAL TRIAL: NCT03681548
Title: A Randomized, Open Label, Two Arm, Single Dose, Crossover, Bioequivalence Study of Ayana Pharma's Doxorubicin Hydrochloride Liposome Injection (LC-101) (Investigational Product) and the US Reference Standard Doxorubicin Hydrochloride Liposome Injection (Sun Pharma), in Subjects With Ovarian Cancer.
Brief Title: A Study of Doxorubicin Hydrochloride Liposome Injection in Subjects With Ovarian Cancer.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ayana Pharma Ltd., (Industry)
Collaborators: Lambda Therapeutic Research Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LC-101-02; 0384-18 (Other: Lambda); CTRI/2018/07/014835 (Registry Identifier: CTRI)
Record Dates: First submitted 2018-09-17; First posted 2018-09-24 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Ovarian Cancer Recurrent
Keywords: liposomal doxorubicin injection; bioequivalence study; ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Intervention Model Description: Bioequivalence study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Reference Product - R (Active Comparator): Doxorubicin Hydrochloride Liposome Injection (Sun Pharma); 20 mg/10 mL i.e. 2 mg/mL (50mg/m2 dose). As this is a cross over study, subjects receiving in Cycle 1 the Reference Product (doxorubicin hydrochloride liposome injection SunPharma), will receive in Cycle 2 the Test Product (doxorubicin hydrochloride liposome injection (Ayana); after at least 4 weeks (RT).
  Interventions: Drug: Doxorubicin Hydrochloride Liposome Injection
- Test Product - T (Experimental): Doxorubicin Hydrochloride Liposome Injection (Ayana Pharma Ltd); 20 mg/10 mL i.e. 2 mg/mL (50mg/m2 dose). As this is a cross over study, subjects receiving in Cycle 1 the Test Product (doxorubicin hydrochloride liposome injection (Ayana)will receive in Cycle 2 the Reference Product (doxorubicin hydrochloride liposome injection SunPharma); after at least 4 weeks (RT).
  Interventions: Drug: Doxorubicin Hydrochloride Liposome Injection

INTERVENTIONS:
Drug: Doxorubicin Hydrochloride Liposome Injection — 50mg/m2, IV on Day 1 of each cycle, On Day 1 of Cycle 1 patients will receive either reference or test product, On Day 1 of Cycle 2 , patients will crossover to the alternate reference or test formulation
  Other Names: Doxorubicin Hydrochloride Liposomal injection 20 mg/10 mL

SUMMARY:
Bioequivalence study is proposed to be carried out on patients of ovarian cancer, who are already receiving or who in the opinion of their treating physicians are candidates for Doxorubicin liposomal injection therapy .

DETAILED DESCRIPTION:
This study is a randomized, open label, two arm, single dose, crossover bioequivalence study. This study will be conducted in female subjects aged 18 to 65 years diagnosed with ovarian cancer whose disease has progressed or recurred after platinum-based chemotherapy and who are already receiving or scheduled to start therapy with Doxorubicin Hydrochloride Liposome Injection product. Each subject will be randomized to one of the two treatment sequences (RT or TR) according to a randomization scheme prepared prior to start of the trial. Serial blood samples for determination of free and liposomal encapsulated doxorubicin plasma concentration for PK analysis will be obtained in each cycle., This study has an adaptive 2-stage design. A sufficient number of subjects with ovarian cancer shall be recruited to have approximately 42 evaluable subjects completing all follow up procedures (Stage 1). An interim analysis of free and encapsulated doxorubicin will be performed at the end of Stage 1. If the bioequivalence of encapsulated and free doxorubicin has been established, then the study will be stopped. Otherwise, the study may continue into Stage 2 with additional number of ovarian cancer subjects. A final evaluation of bioequivalence based on free and encapsulated doxorubicin will be performed at the end of Stage 2 and will include all enrolled subjects completing the study. Bioequivalence criteria: the 94.12% confidence interval of the ratio of geometric means of TEST to REFERENCE for Cmax, AUC0-t, AUC0-∞, for free and encapsulated doxorubicin should be between 80.00% and 125.00%.

ELIGIBILITY:
Inclusion Criteria:

1. Adult female subjects between 18 to 65 years of age (both inclusive) at the time of screening visit.
2. Subjects with histologically or cytological proven ovarian cancer, whose disease has progressed or recurred after platinum-based chemotherapy and scheduled to start therapy with or who are already receiving an approved dose of 50 mg per meter square Doxorubicin Hydrochloride Liposome Injection product.
3. Subjects expected to be able to receive both doses of Doxorubicin Hydrochloride Liposome Injection.
4. Subjects eligible for receiving a dose of 50 mg per meter square of Doxorubicin Hydrochloride Liposome Injection.
5. Subjects with Performance less than or equal to 2 on the Eastern Cooperative Oncology Group (ECOG) performance scale
6. Cardiac function (LVEF) greater than or equal to 50 percentage.
7. Adequate renal, hepatic and bone marrow function without blood product or hematopoietic growth factor support.
8. Subjects able to understand the investigational nature of this study.
9. Availability of subject for the entire study period and willingness to adhere to protocol requirements.
10. For subjects of child-bearing potential, serum beta HCG pregnancy test at screening and urine pregnancy test prior to dosing must be negative and subjects agree to use an acceptable and effective approved method of contraception
11. Subjects of non-childbearing potential who are either surgically sterile (hysterectomy, bilateral oophorectomy, or bilateral tubal ligation) or greater than 1 year postmenopausal with follicle stimulating hormone in the postmenopausal range
12. Signed written informed consent.

Exclusion Criteria:

1. Subjects with history or presence of significant:

   * Allergy or significant history of hypersensitivity or idiosyncratic reactions to a conventional formulation of Doxorubicin Hydrochloride and/or any components of Doxorubicin Hydrochloride liposome injection.
   * Clinically significant pulmonary, hepatic, renal, bone marrow, gastrointestinal, endocrine, immunologic, dermatologic, musculoskeletal, neurological or psychiatric disease.
   * Impaired cardiac function
2. Alcohol dependence, alcohol abuse or drug abuse or addiction with any recreational drug within the past one year.
3. Active opportunistic infection with mycobacteria, cytomegalovirus, toxoplasma, p. carinii or other microorganism (bacterial, viral or fungal).
4. Clinically significant illness (except ovarian cancer) within four weeks prior to dosing.
5. Prior radiation therapy to mediastinum
6. Concomitant use of other cytotoxic or cytostatic drugs or of radiotherapy within four weeks prior to dosing
7. Subject under treatment of myelotoxic drugs, other than doxorubicin (liposomal).
8. Use of prescription or non-prescription herbal and dietary supplements, within 7 days prior to dosing.
9. Subjects with other known active malignancies requiring treatment within 3 years (except for ovarian and/or skin cancer).
10. Subjects with known brain metastasis and/or subjects considered for radiotherapy treatment.
11. Positive result to any of the following: HIV-1/2, hepatitis A, B and C; syphilis.
12. Use of CYP3A4 enzyme-modifying drugs in the previous 30 days prior to dosing and during the study
13. Subjects who have:

    * Systolic blood pressure less than 90 mmHg or more than 160 mmHg
    * Diastolic blood pressure less than 60 mmHg or more than 95 mmHg
    * Pulse rate below 55 per min. or above 100 per min14.
14. Subjects with abnormal laboratory parameters
15. Subject is currently enrolled in, or has not yet completed a period of at least 30 days since ending other investigational device or drug trial(s).
16. Subjects who are legally detained in an official institute.
17. Subjects with prior doxorubicin exposure that would result in a total lifetime exposure of 550 mg per meter square or more after four cycles of treatment.
18. Has any condition that, in the opinion of the investigator, would make participation not be in the best interest (e.g., compromise the well-being) of the subject or that could prevent, limit, or confound the protocol-specified assessments
19. Females of childbearing potential unwilling to use acceptable contraception (as identified in the protocol) throughout the trial and for 6 months after the last dose of study drug.
20. Pregnant or breast-feeding subjects.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-08-29 (Actual); Primary Completion 2019-02-08 (Actual); Study Completion 2019-03-07 (Actual)

PRIMARY OUTCOMES:
Assessment of bioequivalence using Cmax of encapsulated and free doxorubicin in plasma | Throughout 15 days after both dosing.
  Assessment of bioequivalence of LC-101 (TEST Product) in comparison to the US Reference standard (REFERENCE product). Bioequivalence will be assessed using maximum plasma doxorubicin concentration (Cmax) of encapsulated and free doxorubicin measurements in plasma.
Assessment of bioequivalence using AUC (0-t) of encapsulated and free doxorubicin in plasma | Throughout 15 days after both dosing.
  Assessment of bioequivalence of LC-101 (TEST Product) in comparison to the US Reference standard (REFERENCE product). Bioequivalence will be assessed using areas under the plasma concentration versus time curve calculated from 0 to the last measurable observation (AUC 0-t) of encapsulated and free doxorubicin measurements in plasma.
Assessment of bioequivalence using AUC (0-inf) of encapsulated and free doxorubicin in plasma | Throughout 15 days after both dosing.
  Assessment of bioequivalence of LC-101 (TEST Product) in comparison to the US Reference standard (REFERENCE product). Bioequivalence will be assessed using areas under the plasma concentration versus time curve calculated from 0 to infinity (AUC 0-inf) of encapsulated and free doxorubicin measurements in plasma.

SECONDARY OUTCOMES:
Assessment of bioequivalence using Cmax of total doxorubicin in plasma | Throughout 15 days after both dosing.
  Assessment of bioequivalence of LC-101 (TEST Product) in comparison to the US Reference standard (REFERENCE product). Bioequivalence will be assessed using Cmax of total doxorubicin measurements in plasma.
Assessment of bioequivalence using AUC (0-t) of total doxorubicin in plasma | Throughout 15 days after both dosing.
  Assessment of bioequivalence of LC-101 (TEST Product) in comparison to the US Reference standard (REFERENCE product). Bioequivalence will be assessed using AUC (0-t) of total doxorubicin measurements in plasma.
Assessment of bioequivalence using AUC (0-inf) total doxorubicin as secondary analyte | Throughout 15 days after both dosing.
  Assessment of bioequivalence of LC-101 (TEST Product) in comparison to the US Reference standard (REFERENCE product). Bioequivalence will be assessed using AUC (0-inf) of total doxorubicin measurements in plasma.
Assessment of safety | Troughout 42 days after first dosing
  Assessment of incidence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Rakesh J Patel, MD Pharm, Study Director — Lambda Therapeutic Research Ltd.
Locations (15):
- India (15):
  - MNJ Institute of Oncology & Regional Cancer Center, Hyderabad, Andhra Pradesh
  - HCG City Cancer Centre, Vijayawada, Andhra Pradesh
  - Mahatma Gandhi Cancer Hospital & Research Institute, Visakhapatnam, Andhra Pradesh
  - Nirmal Hospital Pvt. Ltd., Surat, Gujarat
  - Unique Hospital - Multispeciality and Research Institute, Surat, Gujarat
  - Aman Hospital and Research Center, Vadodara, Gujarat
  - Kailash Cancer Hospital And Research Center, Vadodara, Gujarat
  - K R Hospital, Mysore, Karnataka
  - Apex Wellness Rishikesh Hospital, Nashik, Maharashtra
  - HCG Manavata Cancer Centre, Nashik, Maharashtra
  - Noble Hospital Pvt Ltd., Pune, Maharashtra
  - Sparsh Hospitals & Critical Care (P) Ltd., Bhubaneshwar, Odisha
  - Sri Ramachandra Medical Centre, Chennai, Tamil Nadu
  - Saveetha Medical College & Hospital, Chennai, Tamil Nadu
  - VGM Hospital, Coimbatore, Tamil Nadu

IPD SHARING:
Plan to Share IPD: No